CLINICAL TRIAL: NCT06414785
Title: INFLAMA : Histological and Molecular Characterization of Capsule Inflammation in Patients Exposed to Silicone Breast Implants
Brief Title: Characterization of Capsule Inflammation in Patients Exposed to Silicone Breast Implants
Acronym: INFLAMA
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Institut de Science des Matériaux de Mulhouse IS2M (Unknown); NOVOTEC labs (lyon) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2024/870
Record Dates: First submitted 2024-05-03; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Breast Implant; Complications; Breast Expansion Prosthesis
Keywords: type of texturing of implants; periprosthetic capsule fragment

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: analysis of samples of periprosthetic capsules taken during breast implant change procedure — characteristics of inflammation and the importance of silicone exposure (intact implant, implant rupture in serum or silicone) at the genomic molecular level, by analyzing the level of expression of genes related to the extracellular matrix and inflammation within a periprosthetic capsule fragment

SUMMARY:
The use of breast implants, both in cosmetic and restorative surgery, is common. It is a device consisting of a silicone elastomer envelope and the container of which may be silicone gel or saline. They can be texturing carriers (roughness) on the surface of their envelope.

If silicone is considered inert and biocompatible, several phenomena should be noted:

* Implant placement results in the formation of a periprosthetic capsule which is the product of the inflammatory reaction and will isolate it from adjacent breast tissue
* The periprosthetic capsule and adjacent breast tissue are chronically exposed to implant silicone.
* Silicone in implants, even intact, has been shown to diffuse through the shell into the periprosthetic compartment and adjacent breast tissue
* There is a phenomenon of erosion of the surface of the implants, particularly textured, responsible for the release of silicone particles within the periprosthetic capsule
* The rupture of the prosthetic envelope is a dreaded complication, due to the alteration of the aesthetic result and the possibility of leakage of silicone gel
* Since 2016, macrotextured implants have been implicated in the occurrence of anaplastic large cell lymphoma associated with breast implants (LAC-AIM) The presence of silicone in contact with tissues seems to promote an inflammatory environment, and this phenomenon seems increased if the implant is textured.

Chronic inflammation induced by these devices can therefore have harmful consequences in the long term. INFLAMA study interested in the consequences of the presence of a silicone implant on local inflammatory phenomena within the periprosthetic capsule.

ELIGIBILITY:
Inclusion Criteria:

* Women over the age of 18 years old
* Requiring a change of unilateral/bilateral breast implants or breast expansion prosthesis for cosmetic surgery or breast reconstruction
* Subject not objecting to the use of personal data and/or biological samples
* Affiliation to or beneficiary of a French social security scheme.

Exclusion Criteria:

* Transgender men and patients
* Pregnant women, and nursing mothers
* Persons deprived of their liberty by a judicial or administrative decision;
* Persons undergoing psychiatric care under duress;
* Persons admitted to a health or social establishment for purposes other than research
* Persons of full age who are subject to a legal protection measure or who cannot express their consent
* Subject being in the period of exclusion from another study or foreseen by the "national volunteer file".

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Women Requiring a change of unilateral/bilateral breast implants or breast expansion prosthesis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-05-03 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
characteristics of inflammation according to the importance of silicone exposure | immediately after surgery
  Verify the existence of a relationship between the characteristics of inflammation and the importance of silicone exposure (intact implant, implant rupture in serum or silicone) at the genomic molecular level, by analyzing the level of expression of genes related to the extracellular matrix and inflammation within a periprosthetic capsule fragment

SECONDARY OUTCOMES:
characteristics of inflammation according to the type of texturing of implants | immediately after surgery
  Check the existence of a relationship between the characteristics of inflammation and the type of texturing of implants (smooth, micro textured or macro textured), on the genomic molecular level, by analyzing the level of expression of genes related to the extracellular matrix and inflammation within a periprosthetic capsule fragment.
Characterize the inflammatory reaction within the periprosthetic capsule histologically, depending on the importance of silicone exposure. | immediately after surgery
Characterize the inflammatory reaction within the periprosthetic capsule histologically, according to texturation. | immediately after surgery
Identify a possible relationship between the characteristics of inflammation and the presence of a clinical shell. | immediately after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle PLUVY, Principal Investigator — CHU de Besançon
Locations (1):
- CHU de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No